CLINICAL TRIAL: NCT01197820
Title: Hepatic and Renal Thermography Using Magnetic Resonance Imaging
Acronym: THeR-IRM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2010/11
Record Dates: First submitted 2010-09-02; First posted 2010-09-09 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Liver Tumors; Kidney Carcinoma
Keywords: HIFU; mobile organs; thermometry; MR; liver; kidney; cancer; Liver tumors, kidney carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): 30 patients with liver tumour and 15 patients with kidney tumour will be enrolled.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Patients will have a regular hepatic or kidney MRI investigation; we will add our sequences on their initial protocol. At first, one thermometry sequence is performed before angular correction is achieved with the following parameters: FOV=300 mm, matrix=96*96, TE/TR=18/72 ms, 67 lines/TR, Sense factor=1.4, 5 slices (4 coronal et 1 sagittal), 30° Flip angle.
  In order to determine the main direction of motion, a set of 200 images are acquired during motion with two interleaved orthogonal slices (one coronal and one sagittal) centered on the region of interest, with the read out direction aligned with the head-feet direction. True-fisp images are acquired during 40 seconds with the following parameters: FOV=400 mm, matrix=128*109, TE/TR=1.2/2.43 ms, 60° flip angle, and 6 mm slice thickness.
  Then the tested software proposes an angular correction to minimize out of plane motion. For each set of orientations, MR thermometry is performed

SUMMARY:
Several technological challenges exist to apply Magnetic Resonance guided High Intensity Focused Ultrasound (MRgHIFU) for treatment of liver or kidney in particular challenges related to the motion of these organs. This study tests a new software to improve thermometry accuracy in mobile organs in patients with liver or kidney tumors. In the same time, the trajectory of the target in 3D is analyzed.

DETAILED DESCRIPTION:
Liver and kidney tumors represent a major health problem because most patients are unsuitable for curative treatment with surgery. Thus, percutaneous ablation, using radio frequency (RF), is preferred : an interstitial electrode that delivers alternative current is placed into the tissue. Consequently, the development of an accurate and completely non-invasive method based on MR guided HIFU treatment is of particular interest since the energy source is located outside the body. There is no incision. For the patient, it provides a treatment option with reduced trauma and improved quality of life, and for the society, it provides reduced hospitalization time and reduced costs.

MRgHIFU has already been tested clinically in tumors of immobilized tissues as uterine leiomyoma. However, several technological challenges exist to apply it for treatment of the liver or the kidney especially challenges related to the motions of these organs. In order to improve the therapeutic efficiency and the safety of the intervention, real time mapping of temperature and thermal dose appear to offer the best strategy to optimize such interventions and provide clinical therapy endpoints. Among imaging modalities, MRI Proton Resonance Frequency based method appears to be the ideal tool for temperature mapping.

One major drawback of PRF thermometry is its high sensitivity to motion. Therefore motion correction is necessary to use PRF thermometry in mobile organs such as the liver or kidneys. To correct artefacts generated in temperature maps by periodical organ motion, a new technique was developed in the IMF lab of Bordeaux University Hospital.

The primary outcome of this study is to evaluate the precision of multiplanar MR imaging with real time motion compensation in hepatic or renal tumour patient.

Secondary outcomes are :

* Characterization of 3d movements of the tumour and test if imaging is improved when the imaging plan contains the main axis of movement.
* Ballistic: we need to identify all anatomical structures which are in the way of the HIFU beam in order to define the types of tumour suitable for future treatments
* Another outcome is to define what modifications are needed in order to treat patients such as depth of treatment, power level. We also need to see the target, ribs, and the transducer in order to evaluate the number of transducer elements to be turned off during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Liver tumors treated or not : HCC, liver metastases of colorectal cancer, hepatocellular adenoma, focal and nodular hyperplasia,
* Kidney tumors : carcinoma
* more than 18 years old

Exclusion Criteria:

* Tumours of the liver dome
* Deprived of their liberty by court
* Pregnant woman
* Contraindication to MRI examination
* Contraindication to including gadolinium salts injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Temperature standard deviation | Duration of MRI specific sequence (15 min)
  To test the ability of this method to improve thermometry accuracy, temperature standard deviations will be studied. Indeed, temperature standard deviations reflect thermometry inaccuracy in absence of temperature variations. Temperature standard deviation in each pixel will be measured over a temporal window. Two regions of interest (ROI) determined by the operator will be considered: the first one in the tumor, the second one for the whole organ.

SECONDARY OUTCOMES:
Characterization of tumor motion in 3D during respiratory cycles | Duration of MRI specific sequence (15 min)
  To characterize tumor motion in the 3 dimensions during respiratory cycles :
  To study the ability of this approach to determinate the 3D trajectory of a target, motion projections on three orthogonal axes will be analyzed from the MRI two orthogonal slices. If the motion can be assimilated to a rectilinear displacement, there will be amplitude minimization after angular correction.
Improve of MRgHIFU shooting ballistics: | Duration of MRI specific sequence (15 min)
  we need to see all anatomical structures in the path of the HIFU cone. Depth of the tumour, number of ribs in the pathway, presence of sensitive organ in the pathway or in PTV vicinity will be recorded
HIFU platform improvements | Duration of MRI specific sequence (15 min)
  To define what improvements are needed on the HIFU platform in order to enhance its therapeutical abilities (depth of treatment, power level…) Amount of transducer's elements masked by rib's shadow, calculation of power level required for treatment, required number of HIFU transducer elements to be turn-off will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé TRILLAUD, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Service de radiologie - Hôpital PELLEGRIN - CHU de Bordeaux, Bordeaux
  - Service of medical Imaging St André Hospital - CHU de BORDEAUX, Bordeaux